CLINICAL TRIAL: NCT02846545
Title: SIMPONI® to Arrest β-cell Loss in Type 1 Diabetes
Brief Title: A Study of SIMPONI® to Arrest Beta-cell Loss in Type 1 Diabetes
Acronym: T1GER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108187; CNTO148DML2001 (Other: Janssen Research & Development, LLC); 2021-000189-13 (EudraCT Number)
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Golimumab (Experimental): Participants will receive subcutaneous (SC) golimumab intermittently for 52 weeks in double-blind period, where doses will be based on weight and/or body surface area. Participants meeting response criteria at Week 52, may enter in an open-label (OL) extension period to receive golimumab SC for 50 weeks (doses will be based on weight and/or body surface area).
  Interventions: Biological: Golimumab
- Group 2: Placebo (Placebo Comparator): Participants will receive a matching placebo to golimumab.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Golimumab — Participants will receive subcutaneous golimumab intermittently for 52 weeks in double-blind period, where doses will be based on weight and/or body surface area. Participants meeting response criteria at Week 52, may receive golimumab SC for 50 weeks (doses will be based on weight and/or body surface area) in an OL extension period.
  Other Names: SIMPONI
  Arms: Group 1: Golimumab
Biological: Placebo — Matching Placebo to golimumab.
  Arms: Group 2: Placebo

SUMMARY:
The primary purpose of this study is to determine if golimumab can preserve beta-cell function in children and young adults with newly diagnosed Type 1 Diabetes (T1D).

ELIGIBILITY:
Inclusion Criteria:

Double-blind Period:

* Be positive for at least 1 of the following diabetes-related autoantibodies obtained at study screening: Glutamic acid decarboxylase (GAD-65), islet antigen 2 (IA-2), zinc transporter 8 (ZnT8), Islet Cell Cytoplasmic Autoantibodies (ICA), or Insulin (if obtained within 10 days of the onset of exogenous insulin therapy)
* Have a peak stimulated C-peptide level greater than or equal to (>=) 0.2 picomole per milliliter (pmol/mL) following a 4-hour Mixed-meal Tolerance Test (MMTT) obtained at study screening
* Be medically stable on the basis of physical examination, medical history, and vital signs performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population
* Females of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) test at screening and a negative urine pregnancy test at the Week 0 visit
* Participants (or their legally acceptable representatives) are willing and able to adhere to requirements, prohibitions, and restrictions specified in this protocol

Open-Label Extension Period:

- Participants must meet the responder criteria based on C-peptide area under the concentration-time curve (AUC) and insulin dose-adjusted HbA1c (IDAAC) remission score

Exclusion Criteria:

Double-blind Period:

* Has a history of significant renal, vascular, pulmonary, gastrointestinal, neurologic, hematologic, rheumatologic, or psychiatric disease or immune suppression or immune deficiency.
* Has significant cardiovascular disease, including history of myocardial infarction, congestive heart failure, angina, abnormal electrocardiogram or abnormal stress test
* Has active infections, is prone to infections or has chronic, recurrent or opportunistic infectious disease, including but not limited to, chronic renal infection, chronic chest infection (example [eg.], bronchiectasis), sinusitis, recurrent urinary tract infection (eg., recurrent pyelonephritis, chronic cystitis), Pneumocystis carinii, aspergillosis, latent or active granulomatous infection, histoplasmosis, or coccidioidomycosis or an open, draining, or infected non-healing skin wound or ulcer
* Has a clinically active infection with Epstein-Barr virus (EBV) or an EBV viral load >=10,000 copies per milliliter (mL) of plasma obtained at study screening. Has a clinically active infection with cytomegalovirus (CMV) or a CMV viral load >= 10,000 copies per milliliter (mL) of plasma obtained at study screening
* Current or prior (within 30 days of screening) treatment that is known to cause a significant, ongoing change in the course of T1D or immunologic status, including high-dose inhaled, extensive topical, or systemic glucocorticoids
* Has another autoimmune disease (eg, rheumatoid arthritis [RA], polyarticular juvenile idiopathic arthritis [pJIA], psoriatic arthritis [PsA], ankylosing spondylitis [AS], multiple sclerosis [MS], systemic lupus erythematosus [SLE], celiac disease [clinically symptomatic and antibody positive, that is, tissue transglutaminase Immunoglobulin A [IgA]) excluding clinically stable autoimmune thyroiditis whether treated or untreated
* Has any of the following tuberculosis [TB] screening criteria: A history of latent or active TB prior to screening (including but not limited to a positive QuantiFERON®-TB Gold test), signs or symptoms suggestive of active TB upon medical history and/or physical examination, recent close contact with a person with known or suspected active TB
* Has known allergies, intolerance and/or hypersensitivity to human immunoglobulin proteins, golimumab or any of its components or its excipients

Open-Label Extension Period:

* Participants having reported clinically significant AEs or serious adverse events (SAEs) deemed to be related to the study agent during the double blind period (for example. severe infections or hypersensitivity reactions), precluding renewed exposure to golimumab
* Participants who discontinued study agent administration prior to Week 52 or who have completed the Week 104 visit of the double-blind period or discontinued early from study

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (33):
- United States (33):
  - Little Rock, Arkansas
  - Newport Beach, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Walnut Creek, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Doral, Florida
  - Gainesville, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Morristown, New Jersey
  - Buffalo, New York
  - The Bronx, New York
  - Mentor, Ohio
  - Philadelphia, Pennsylvania
  - Sioux Falls, South Dakota
  - Dallas, Texas
  - San Antonio, Texas
  - Schertz, Texas
  - Webster, Texas
  - Seattle, Washington
  - Tacoma, Washington

REFERENCES:
- [Derived] Quattrin T, Haller MJ, Steck AK, Felner EI, Li Y, Xia Y, Leu JH, Zoka R, Hedrick JA, Rigby MR, Vercruysse F; T1GER Study Investigators. Golimumab and Beta-Cell Function in Youth with New-Onset Type 1 Diabetes. N Engl J Med. 2020 Nov 19;383(21):2007-2017. doi: 10.1056/NEJMoa2006136. PMID 33207093

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants in the active treatment period received a subcutaneous (SC) injection of placebo every 2 weeks (q2w) from Week (Wk) 0 through Week 52 to match the active arm. Following the 52-week active treatment period, participants were monitored for an additional 52 weeks for safety (off-therapy follow-up [FU] period).
- Golimumab: Participants in active treatment period weighing less than (<) 45 kilograms (kg) received an induction dose of golimumab 60 milligrams/ meter square (mg/m^2) SC injection at Weeks 0 and 2 followed by a maintenance dose of golimumab 30 mg/m^2 SC injection at Week 4 and q2w through Week 52. Participants weighing greater than and equal to (>=45) kg received an induction dose of golimumab 100 mg SC injection at Weeks 0 and 2 followed by a maintenance dose of golimumab 50 mg SC injection at Week 4 and q2w through Week 52. Following 52-week active treatment period, participants were monitored for an additional 52 weeks for safety and did not receive study drug during this period (off-therapy follow-up period). Participants were assessed for response at Week 52 and those who were responders and still in the off-therapy follow-up period were offered option to enter open-label extension (OLE) period after active treatment period, if eligibility criteria were met. Participants weighing <45 kg received a maintenance dose of golimumab 30 mg/m^2 SC injection at Week 0 and q2w thereafter through OLE Week 52. Participants weighing >=45 kg received maintenance dose of golimumab 50 mg/m^2 SC injection at Week 0 and q2w thereafter through OLE Week 52. After OLE Week 52, participants were followed up for safety up to OLE Week 60. Non-responders at Week 52 continued in off-therapy follow-up period in which they were monitored for safety for additional 52 weeks and did not receive study drug.
Period: Active Treatment Period: Week 0-52
Arm/Group | Placebo | Golimumab
Started | 28 | 56
Completed | 25 | 50
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5
Period: Off-therapy FU:Wk 52-104 & OLE: Wk 0-60
Arm/Group | Placebo | Golimumab
Started | 25 | 49 (1 participant from the golimumab treatment group terminated study participation on the day of the Week 52 visit.)
Participants Who Entered OLE Period | 0 | 5
Participants Who Completed OLE Period | 0 | 1
Completed | 23 | 47
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Golimumab | Total
Number analyzed (Participants) | 28 | 56 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (4.01) | 13.3 (3.73) | 13.4 (3.8)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 8 | 20 | 28
  Adolescents (12-17 years) | 13 | 27 | 40
  Adults (18-64 years) | 7 | 9 | 16
  From 65 to 84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 25 | 35
  Male | 18 | 31 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 26 | 51 | 77
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 26 | 46 | 72
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Active Treatment Period: C-peptide Area Under the Concentration-time Curve (AUC) Calculated From a 4 Hour Mixed Meal Tolerance Test (MMTT) at Week 52
Description: MMTT-Stimulated 4-Hour C-peptide AUC was defined as the mean area under the C-peptide level time curve over the 4-hour period divided by the duration after a mixed-meal tolerance test.
Time Frame: Week 52
Population: Full Analysis Set (FAS) included all randomized participants who took at least one dose (complete or partial) of study agent. Here 'N' (number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: picomoles per milliliter (pmol/mL)
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 25 | 50
picomoles per milliliter (pmol/mL) | 0.43 (0.388) [lower limit 0.388] | 0.64 (0.423) [lower limit 0.423]

2. Secondary Outcome: Active Treatment Period: Change From Baseline in Insulin Use in Units Per Kilogram Body Weight Per Day
Description: Change from baseline in daily insulin use at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: FAS included all randomized participants who took at least one dose (complete or partial) of study agent. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units/kilogram/day
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 17 | 42
units/kilogram/day | 0.239 (0.2225) | 0.057 (0.2850)
Statistical Analysis 1: Comparison: Placebo vs Golimumab; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Least Square (LS) Mean = -0.178, 95% CI 2-sided [-0.28 to -0.08]

3. Secondary Outcome: Active Treatment Period: Change From Baseline in Glycosylated Haemoglobin (HbA1c) at Week 52
Description: Change from baseline in glycosylated HbA1c at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: HbA1C percent (%)
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 28 | 50
HbA1C percent (%) | 0.61 (1.368) | 0.35 (1.851)
Statistical Analysis 1: Comparison: Placebo vs Golimumab; Test type: Superiority; p = 0.8020, Mixed Models Analysis; LS Mean = -0.09, 95% CI 2-sided [-0.81 to 0.63]

4. Secondary Outcome: Hypoglycemic Event Rates
Description: A hypoglycemic event was defined as either a biochemically confirmed hypoglycemic episode or a severe hypoglycemic event. The hypoglycemia event rate (number of hypoglycemia episodes per patient-year) was defined as blood glucose levels of less than and equal to (<=) 70, 55, and 35 mg/dL or clinical sequelae consistent with severe hypoglycemia in the absence of a BG reading.
Time Frame: Up to Week 52
Population: FAS which had all randomized participants who took at least one dose (complete or partial) of study agent.
Measure: Number; unit: events per patient-year
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 28 | 56
events per patient-year | 43.36 | 39.01
Statistical Analysis 1: Comparison: Placebo vs Golimumab; Hypoglycemia rate was analyzed by using a Poisson regression model with the number of hypoglycemia events through Week 52 as the response, treatment and gender as fixed factors, age and baseline HbA1c as covariates, and the duration of study participation through week 52 in logarithm as an offset variable; Test type: Superiority; p = 0.0036, Poisson regression model; Ratio of hypoglycemia rates = 0.90, 95% CI 2-sided [0.838 to 0.966]

5. Secondary Outcome: Active Treatment Period: C-peptide Area Under the Concentration-time Curve (AUC) Calculated From a 4 Hour Mixed Meal Tolerance Test (MMTT) Over Time
Description: MMTT-Stimulated 4-Hour C-peptide AUC is the mean area under the C-peptide level-time curve over the 4-hour period divided by the duration after a mixed-meal tolerance test.
Time Frame: Baseline, Weeks 12, 26, 38, 52, 78 and 104
Population: FAS included all randomized participants who took at least one dose (complete or partial) of study agent. Here 'n' (number analyzed) included all participants who were analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 28 | 56
pmol/mL
  Baseline | 0.88 (0.634) | 0.78 (0.396)
  Week 12: number analyzed (Participants) | 26 | 52
  Week 12 | 0.62 (0.426) | 0.78 (0.355)
  Week 26: number analyzed (Participants) | 25 | 49
  Week 26 | 0.55 (0.424) | 0.76 (0.380)
  Week 38: number analyzed (Participants) | 24 | 49
  Week 38 | 0.53 (0.423) | 0.73 (0.424)
  Week 52: number analyzed (Participants) | 25 | 50
  Week 52 | 0.43 (0.388) | 0.64 (0.423)
  Week 78: number analyzed (Participants) | 24 | 47
  Week 78 | 0.31 (0.264) | 0.45 (0.385)
  Week 104: number analyzed (Participants) | 21 | 40
  Week 104 | 0.25 (0.273) | 0.35 (0.360)

6. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability
Description: An adverse event (AE) was defined as any untoward medical occurrence in clinical study subject administered medicinal product. It could be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. Treatment emergent AEs were defined as AEs with onset during the treatment phase or that are a consequence of a pre-existing condition that has worsened since baseline.
Time Frame: Up to Week 52 (Active treatment period), Up to Week 104 (Active treatment + Off therapy follow-up period)
Population: The safety analysis set included all randomized participants who received at least 1 (partial or complete) dose of study agent, that is, the treated population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 28 | 56
percentage of participants
  Up to Week 52 | 82.1 | 91.1
  Up to Week 104 | 89.3 | 96.4

7. Secondary Outcome: Percentage of Participants With Serious Adverse Events
Description: An AE was defined as any untoward medical occurrence in clinical study participant administered medicinal product. It could be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. A serious AE was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious treatment via medicinal product and was medically important.
Time Frame: Up to Week 52 (Active treatment period), Up to Week 104 (Active treatment + Off therapy follow-up period)
Population: as for outcome 6
Measure: Number; unit: percentage participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 28 | 56
percentage participants
  Up to Week 52 | 3.6 | 1.8
  Up to Week 104 | 7.1 | 8.9

8. Secondary Outcome: Percentage of Participants With Severe Infections Through Week 52 and Week 104
Description: Participants having 1 or more severe infections were evaluated and reported.
Time Frame: Up to Week 52 (Active treatment period), Up to Week 104 (Active treatment + Off therapy follow-up period)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 28 | 56
percentage of participants
  Up to Week 52 | 60.7 | 71.4
  Up to Week 104 | 67.9 | 75.0

9. Secondary Outcome: Active Treatment Period: Percentage of Participants With Study Agent Injection Site Reactions Up to Week 52
Description: Percentage of participants with study agent injection site reactions up to Week 52 were reported.
Time Frame: Up to Week 52
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 28 | 56
percentage of participants | 28.6 | 23.2

10. Secondary Outcome: Serum Golimumab Concentrations
Description: Serum samples were collected for the measurement of golimumab concentrations.
Time Frame: Preinjection: Week 0, Week 2, Week 4, Week 8, Week 12, and Week 26, Week 33, Week 38 (preinjection),Week 45 and Week 52 (preinjection), for active treatment period; Weeks 78 and 104 for Off-therapy follow-up period
Population: PK Analysis Set included all participants who received at least 1 golimumab injection and had sufficient PK samples for analysis. Here 'n' (number analyzed) included all participants who were analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Golimumab
Number analyzed (Participants) | 56
micrograms per milliliter (mcg/mL)
  Week 0 | 0.00 (0.000)
  Week 2 | 4.64 (1.506)
  Week 4 | 6.85 (2.168)
  Week 8: number analyzed (Participants) | 54
  Week 8 | 4.67 (1.930)
  Week 12: number analyzed (Participants) | 52
  Week 12 | 3.74 (2.032)
  Week 26: number analyzed (Participants) | 50
  Week 26 | 3.37 (2.011)
  Week 33: number analyzed (Participants) | 49
  Week 33 | 4.41 (2.825)
  Week 38: number analyzed (Participants) | 50
  Week 38 | 3.06 (2.127)
  Week 45: number analyzed (Participants) | 49
  Week 45 | 4.44 (2.828)
  Week 52: number analyzed (Participants) | 49
  Week 52 | 2.89 (2.022)
  Week 78: number analyzed (Participants) | 47
  Week 78 | 0.00 (0.007)
  Week 104: number analyzed (Participants) | 38
  Week 104 | 0.00 (0.000)

11. Secondary Outcome: Number of Participants With Antibodies to Golimumab
Description: Number of participants with antibodies to golimumab were reported.
Time Frame: Up to Week 52 (Active treatment period), Up to Week 104 (Active treatment + Off therapy follow-up period)
Population: PK Analysis Set included all participants with appropriate samples (had 1 or more samples) obtained after their first study agent administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab
Number analyzed (Participants) | 56
Participants
  Up to Week 52 | 30
  Up to Week 104 | 37

12. Secondary Outcome: Titers of Antibodies to Golimumab
Description: Titers of antibodies to golimumab were evaluated.
Time Frame: Up to Week 52 (Active treatment period), Up to Week 104 (Active treatment + Off therapy follow-up period)
Population: PK Analysis Set included all the participants who were antibody positive, the peak titers for them were evaluated. Data was not collected and analyzed for this outcome measure due to change in planned analysis.
Arm/Group | Golimumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to Week 52 (Active treatment period), From Week 52-104 (Off-therapy follow-up period), Open label extension (OLE) Week 0-60 after active treatment period (OLE period)
Description: The safety analysis set included all randomized participants who received at least 1 (partial or complete) dose of study agent.
Groups:
- Active Treatment Period: Placebo (Week 0 - 52): Participants in the active treatment period received a subcutaneous (SC) injection of placebo every 2 weeks (q2w) from Week 0 through Week 52 to match the active arm.
- Active Treatment Period: Golimumab (Week 0 - 52): Participants in the active treatment period weighing less than (<) 45 kilograms (kg) received an induction dose of golimumab 60 milligrams/ meter square (mg/m^2) SC injection at Weeks 0 and 2 followed by a maintenance dose of golimumab 30 mg/m^2 SC injection at Week 4 and q2w through Week 52. Participants weighing greater than and equal to (>=45) kg received an induction dose of golimumab 100 mg SC injection at Weeks 0 and 2 followed by a maintenance dose of golimumab 50 mg SC injection at Week 4 and q2w through Week 52.
- Off-therapy Follow Up Period: Placebo (Week 52 - 104): Following the 52-week active treatment period, participants were monitored for an additional 52 weeks for safety (off-therapy follow-up period).
- Off-therapy Period: Golimumab (Week 52 - 104): Following the 52-week active treatment period, participants were monitored for an additional 52 weeks for safety (off-therapy follow-up period) and did not receive the study drug during this period (off-therapy follow-up period).
- OLE Period: Golimumab (OLE Week 0-60 After Active Treatment Period): Following the active treatment period, participants were assessed for response at Week 52 and and those who were responders and still in the off-therapy follow-up period were offered the option to enter the open-label extension (OLE) period. Participants weighing <45 kg received a maintenance dose of golimumab 30 mg/m^2 SC injection at Week 0 and q2w thereafter through OLE Week 52. Participants weighing >=45 kg received maintenance dose of golimumab 50 mg/m^2 SC injection at Week 0 and q2w thereafter through OLE Week 52. After OLE Week 52, participants were followed up for safety up to OLE Week 60. Non-responders at Week 52 continued in the off-therapy follow-up period in which they were monitored for safety for additional 52 weeks and did not receive study drug.
Arm/Group | Active Treatment Period: Placebo (Week 0 - 52) | Active Treatment Period: Golimumab (Week 0 - 52) | Off-therapy Follow Up Period: Placebo (Week 52 - 104) | Off-therapy Period: Golimumab (Week 52 - 104) | OLE Period: Golimumab (OLE Week 0-60 After Active Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/56 | 0/25 | 0/49 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/56 | 1/25 | 4/49 | 1/5
Other Adverse Events (participants affected / at risk) | 21/28 | 45/56 | 14/25 | 26/49 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment Period: Placebo (Week 0 - 52) (N=28) | Active Treatment Period: Golimumab (Week 0 - 52) (N=56) | Off-therapy Follow Up Period: Placebo (Week 52 - 104) (N=25) | Off-therapy Period: Golimumab (Week 52 - 104) (N=49) | OLE Period: Golimumab (OLE Week 0-60 After Active Treatment Period) (N=5)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment Period: Placebo (Week 0 - 52) (N=28) | Active Treatment Period: Golimumab (Week 0 - 52) (N=56) | Off-therapy Follow Up Period: Placebo (Week 52 - 104) (N=25) | Off-therapy Period: Golimumab (Week 52 - 104) (N=49) | OLE Period: Golimumab (OLE Week 0-60 After Active Treatment Period) (N=5)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (7) | 1 (1) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0) | 4 (5) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 3 (4) | 9 (36) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 2 (2) | 6 (11) | 0 (0) | 0 (0) | 0 (0)
Injection Site Swelling (General disorders) | 0 (0) | 4 (14) | 0 (0) | 0 (0) | 0 (0)
Injection Site Urticaria (General disorders) | 3 (13) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (5) | 0 (0) | 2 (2) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 6 (6) | 2 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (8) | 10 (16) | 3 (4) | 4 (5) | 1 (1)
Otitis Media (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (11) | 17 (31) | 4 (4) | 8 (9) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Glycosylated Haemoglobin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (63) | 14 (104) | 2 (90) | 9 (141) | 2 (9)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 11 (27) | 1 (1) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 9 (10) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (9) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT02846545/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT02846545/SAP_001.pdf